CLINICAL TRIAL: NCT07259538
Title: A Phase I Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of VVN432 Nasal Spray in Healthy Chinese Adult Subjects and Patients With Chronic Rhinosinusitis.
Brief Title: A Phase I Study Evaluating the Safety, Tolerability, and Pharmacokinetics of VVN432 Nasal Spray
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: VivaVision Biotech, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VVN432-CCS-101
Record Dates: First submitted 2025-11-16; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Chronic Rhinosinusitis (CRS)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Part 1: 0.5% VVN432 Nasal Spray (1 spray/nostril) (Experimental): 0.5% VVN432 Nasal Spray, single dose, 1 spray/nostril
  Interventions: Drug: 0.5% VVN432 Nasal Spray
- Part 1: 1% VVN432 Nasal Spray (1 spray/nostril) (Experimental): 1% VVN432 Nasal Spray, single dose, 1 spray/nostril
  Interventions: Drug: 1% VVN432 Nasal Spray
- Part 1: 1% VVN432 Nasal Spray (2 spray/nostril) (Experimental): 1% VVN432 Nasal Spray, single dose, 2 sprays/nostril
  Interventions: Drug: 1% VVN432 Nasal Spray
- Part 1: Vehicle (Placebo Comparator): VVN432 Nasal Spray Placebo, single dose, 1 or 2 sprays/nostril
  Interventions: Drug: Vehicle
- Part 2: 0.5% VVN432 Nasal Spray (1 spray/nostril) (Experimental): 0.5% VVN432 Nasal Spray, BID, 1 spray/nostril, for 28 days
  Interventions: Drug: 0.5% VVN432 Nasal Spray
- Part 2: 1% VVN432 Nasal Spray (1 spray/nostril) (Experimental): 1% VVN432 Nasal Spray, BID, 1 spray/nostril, for 28 days
  Interventions: Drug: 1% VVN432 Nasal Spray
- Part 2: 1% VVN432 Nasal Spray (2 sprays/nostril) (Experimental): 1% VVN432 Nasal Spray, BID, 2 sprays/nostril, for 28 days
  Interventions: Drug: 1% VVN432 Nasal Spray
- Part 2: Vehicle (Placebo Comparator): VVN432 Nasal Spray Placebo, BID, 1 or 2 sprays/nostril, for 28 days
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: 0.5% VVN432 Nasal Spray — 0.5% VVN432 Nasal Spray
  Arms: Part 1: 0.5% VVN432 Nasal Spray (1 spray/nostril); Part 2: 0.5% VVN432 Nasal Spray (1 spray/nostril)
Drug: 1% VVN432 Nasal Spray — 1% VVN432 Nasal Spray
  Arms: Part 1: 1% VVN432 Nasal Spray (1 spray/nostril); Part 1: 1% VVN432 Nasal Spray (2 spray/nostril); Part 2: 1% VVN432 Nasal Spray (1 spray/nostril); Part 2: 1% VVN432 Nasal Spray (2 sprays/nostril)
Drug: Vehicle — VVN432 Nasal Spray, Placebo
  Arms: Part 1: Vehicle; Part 2: Vehicle

SUMMARY:
The goal of this clinical study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of VVN432 Nasal Spray in healthy volunteers (Phase Ia) and in patients with chronic rhinosinusitis (Phase 1b).

This study consists of two parts (Phase 1a and Phase 1b):

Phase 1a (SAD) is a single-center, randomized, double-masked, vehicle-controlled study to assess the safety, tolerability, and PK of VVN432 Nasal Spray in healthy adult subjects.

Phase 1b (MAD) is a multi-center, randomized, double-masked, vehicle-controlled study to assess the safety, tolerability, PK/PD, and preliminary efficacy of VVN432 Nasal Spray in patients with chronic rhinosinusitis.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Healthy male or female subjects aged 18 to 55 years old (inclusive);
* Body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females; body mass index (BMI) within the range of 18.5 to 28.0 kg/m2 (inclusive);
* No clinically significant abnormalities at screening or baseline.

Part 2:

* Male or female patients aged 18 to 55 years old (inclusive);
* Clinically confirmed diagnosis of chronic rhinosinusitis with or without nasal polyps;
* Presence of the following symptoms for >4 weeks before screening: nasal obstruction, mucous or mucopurulent rhinorrhea, facial pain/pressure, and reduced or lost sense of smell;
* Modified Lund-Kennedy (MLK) score ≥ 2 in each nostril by nasal endoscopy;
* Lund-Mackay score (LMK) ≥ 2 in each nostril by CT scan;
* Nasal Construction Score (NCS) ≥ 2.

Exclusion Criteria:

Part 1:

* Known hypersensitivity or contraindications to the study drug or its components;
* History or current conditions that affect the safety or absorption of the investigational drug;
* History of drug abuse or drug dependence;
* Participation in any other clinical trials and receiving an investigational drug within 12 weeks before screening or 5 half-lives, whichever is longer;
* If female, is pregnant or lactating, or intends to become pregnant during the study period.

Part 2:

* Known hypersensitivity or contraindications to the study drug or its components;
* Use of prohibited medications prior to screening and during the course of the study; History of drug abuse or drug dependence;
* Participation in any other clinical trials and receiving an investigational drug within 12 weeks before screening or 5 half-lives, whichever is longer;
* If female, is pregnant or lactating, or intends to become pregnant during the study period.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: To evaluate the safety and tolerability of VVN432 Nasal Spray. | Baseline to Day 10
  Incidence of the AEs and SAEs; change from baseline in laboratory tests, ECG, and vital signs
Part 2: To evaluate the safety and tolerability of VVN432 Nasal Spray | Baseline to Day 35
  Incidence of the AEs and SAEs; change from baseline in laboratory tests, ECT, and vital signs

SECONDARY OUTCOMES:
Part 1: To evaluate the systemic PK of VVN432 Nasal Spray | 48 hours
  Plasma concentration of VVN432, and assess the PK parameters if applicable
Part 1: To evaluate the local PK of VVN432 Nasal Spray | 48 hours
  Local concentration of VVN432 in the eluent of oropharyngeal swabs and nasal swabs, and in nasal lavage fluid post-dose
Part 2: To evaluate the systemic PK of VVN432 Nasal Spray | Day 1, Day 28, and Day 35
  Plasma concentration of VVN432, and assess the PK parameters if applicable
Part 2: To evaluate the local PK of VVN432 Nasal Spray | Day 1, Day 28, and Day 35
  Local concentration of VVN432 in the eluent of nasal swabs post-dose
Part 2: Efficacy: Nasal Congestion Score (NCS) | Baseline to Day 35
  Change from baseline in NCS (0-3, higher scores indicate more severe symptoms)
Part 2: Efficacy: Total Symptom Score (TSS) | Baseline to Day 35
  Change from Baseline in TSS (0-9 [sum of NCS, loss of smell, and average of anterior and posterior rhinorrhea], higher scores indicate more severe symptoms)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Toren Hospital, Beijing, China